CLINICAL TRIAL: NCT01061008
Title: The Effects of Progressive Handgrip Exercise Training on Arteriovenous Fistula Maturation in Chronic Kidney Disease
Brief Title: Handgrip Exercise for Arteriovenous Fistula Maturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangor University (Other)
Collaborators: Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REC No : 07/WNo01/4; Macdonald 07/4 (Other: R & D Reference No)
Record Dates: First submitted 2010-01-22; First posted 2010-02-02 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Kidney Disease
Keywords: Exercise; arteriovenous fistula; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Arteriovenous Fistula | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Handgrip exercise (Experimental): Handgrip exercise - patients allocated to this intervention will carry out an eight week post operative progressive handgrip exercise training program
  Interventions: Other: Post operative progressive handgrip exercise
- Treatment as usual (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Post operative progressive handgrip exercise — As soon as possible post operation the patient will commence an eight week progressive handgrip training intervention
  Arms: Handgrip exercise
Other: Treatment as usual — Continue routine care, with removal of exercise information given to patients(if anye.g. do not give out squeeze balls)
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to investigate whether post operative progressive forearm exercise is effective in improving arteriovenous fistula maturation in chronic kidney disease patients.

DETAILED DESCRIPTION:
The arteriovenous fistula is considered to be the gold standard form of access for haemodialysis patients, however only 37% of haemodialysis patients have this form of access. A possible explanation for this could be the high fistula failure rate due to the lack of maturation. Therefore interventions aimed at enhancing fistula maturation are warranted. One such intervention could be forearm exercise, however this recommendation is not evidence based. Therefore, the purpose of this study is to investigate whether a program of post operative progressive hand grip exercise can improve fistula maturation.

ELIGIBILITY:
Inclusion Criteria:

* Stage 4-5 chronic kidney disease, attending for arteriovenous fistula creation in forearm

Exclusion Criteria:

* Are under the age of 18years;
* Not able to exercise forearm safely (as decided by the patients consultant)
* Have any other uncontrolled medical condition
* Unable to withstand transiently raised systolic blood pressure by 35 mmHg and diastolic by 25 mmHg
* Or are unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Renal unit, Ysbyty Gwynedd, North West Wales NHS Trust, Bangor, Gwynedd, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with stage four and five CKD attending two renal units in North Wales, UK were invited to participate in the study.
Period: Overall Study
Arm/Group | Handgrip Exercise | Treatment as Usual
Started | 16 | 15
Completed | 10 | 9
Not Completed | 6 | 6
Not completed — Badiocephalic fistula failed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Unable to exercise following surgery | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Handgrip Exercise | Treatment as Usual | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (14) | 60 (11) | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Venous Diameter.
Description: Measurements were made using duplex ultrasonagraphy. Measurements were made at predetermined distances 5 to 10 cm proximal to the anastomosis (dependent on wound dressings and turbulent flow around the anastomosis). The scanning position for each patient was traced using transparent sheets which allowed analogous measurement positions for all scans. Cross sectional vascular diameter measurements were made using conventional grey scale B Mode imaging. Diameters were measured from the inner edges of the vascular wall (Wiese & Nonnast-Daniel, 2004).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Handgrip Exercise | Treatment as Usual
Number analyzed (Participants) | 10 | 9
mm | 5.78 (0.51) | 6.42 (0.89)

2. Secondary Outcome: Maximum Handgrip Strength
Time Frame: 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Handgrip Endurance
Time Frame: 3 months
Reporting Status: Not Posted

4. Secondary Outcome: Forearm Muscle Cross Sectional Area
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Including joint, muscle or wound pain was recorded by the patient and also collected actively by the researcher during each weekly phone call to the patient. Other unexpected and serious (fatal, life threatening, or resulted in hospitalization) harms were collected passively as they occurred and during the trial period only.
Arm/Group | Handgrip Exercise | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 2/10 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Handgrip Exercise (N=10) | Treatment as Usual (N=9)
Pain (Surgical and medical procedures) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes